CLINICAL TRIAL: NCT02662673
Title: Evaluation of Focal Treatments of Localized Prostate Cancers With High Intensity Focused Ultrasound Using the Focal One® Device
Acronym: IDITOP-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-817
Record Dates: First submitted 2016-01-18; First posted 2016-01-25 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Localized Prostate Cancer
Keywords: HIFU; Prostate Cancer; Focal; Quality of life; Index study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Localized prostate cancer, Focal treatment. (Other)
  Interventions: Device: Focal High Intensity Focused Ultrasound (HIFU) treatment

INTERVENTIONS:
Device: Focal High Intensity Focused Ultrasound (HIFU) treatment — Focal High Intensity Focused Ultrasound (HIFU) treatment for localized prostate cancer (maximum two foci). HIFU treatment is using high energy ultrasound focused at the focal point to achieve precise tissue destruction. This mini-invasive therapy is using an endo-rectal approach to deliver the treatment, using a probe composed of a combined imaging and treatment transducer. The treatment is monitored by real-time ultrasound. The treatment planning is performed by the urologist, contouring the area to be treated (MRI target + security margins around the tumor) and the treatment phase is automatically performed by the robotic device.

SUMMARY:
Focal treatment of localized prostate cancer aims to destroy the cancerous foci without damaging surrounding tissues to avoid the side effects of radical treatments. This is why focal treatment is positioned as an alternative to radical surgery as well as an alternative to active surveillance.

This study is a feasibility study. It aims at treating the index tumor (the most aggressive one) which determines the vital prognosis of patient, while preserving the maximum surrounding prostatic tissue to preserve quality of life. The expected result is the total destruction of aggressive tumor areas by focal or multifocal treatment strategy using the Focal One® device (EDAP-TMS, Vaulx-en-Velin, France). The tumor destruction is validated by the negative biopsy rate between 6 and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 80 years (inclusive) with a life expectancy of more than 5 years.
* PSA ≤ 10 ng / mL.
* Initial diagnosis of localized prostate cancer (stage T1 or T2).
* Diagnosis confirmed by a multiparametric MRI and subsequent systematic and targeted prostate biopsies (at least 12 sextant biopsies and two biopsies per MRI target).
* Identification of a primary cancer site (index tumor) possibly associated with a second independent tumor (accessory tumor), provided that these tumors are separated by a sextant or the median line.
* Maximum two cancer foci, each one fulfilling the following conditions
* Gleason score of 6 AND biopsy invasion length ≥5 mm,
* OR Gleason score of 6 AND corresponding focal lesion on MRI with a PIRADS (Prostate Imaging Reporting and Data System) score ≥4/5 and a diameter ≥5 mm,
* OR Gleason score of 7 (3+4) whatever the biopsy invasion length or the MRI results may be.
* Patient with normal anal and rectal anatomy.
* Patient with a condition corresponding to an ASA (American Society of Anesthesiologists) classification 1 or 2.
* Patient for which treatment by focal HIFU (without performing an associated TURP) has been validated in Multidisciplinary meeting.
* Accepting patient monitoring constraints defined in the context of the study.
* Patient affiliated to health insurance or beneficiary a similar plan.

Exclusion Criteria:

* Patient with ASA (American Society of Anesthesiologists) score 3.
* Patient clinical stage T3.
* Metastatic or distant (CT and/or MRI) lymph node.
* Patient with more than two cancer foci.
* Patients already treated for his prostate cancer (hormone therapy, radiotherapy, surgery).
* Patient having a distance between the rectal mucosa and the prostatic capsule over 8 mm.
* History of inflammatory bowel disease, rectal or urinary tract fistula.
* History of pelvic radiotherapy.
* History of bladder cancer.
* History of sclerosis of the bladder neck or urethral stricture.
* Patient with an implant located at least 1 cm of the treatment zone (stent, catheter).
* Hemorrhagic risk patient.
* Urogenital infection in progress.
* Latex allergy.
* Allergy to sulfur hexafluoride or any of the other components of SonoVue®.
* Patients with recent acute coronary syndrome or unstable ischemic heart disease: myocardial infarction phase formation or evolution, typical angina at rest within last 7 days, significant worsening of cardiac symptoms within last 7 days, recent intervention on the coronary arteries or other factors suggesting clinical instability (eg recent ECG changes, changes in clinical or laboratory parameters), acute heart failure, heart failure stage III or IV, or severe rhythm disorders (contra-indications to the use of SonoVue®).
* Patient with a right to left shunt, severe pulmonary hypertension (pulmonary artery pressure> 90 mm Hg), uncontrolled systemic hypertension.
* Patient with respiratory distress syndrome.
* Patient with severe chronic obstructive pulmonary disease.
* Patient with acute endocarditis, prosthetic valve holder, acute systemic inflammation and / or sepsis, hyper coagulation status and / or recent thromboembolism.
* Patient on life support or suffering from unstable neurological diseases.
* Contra-indication for MRI (pacemakers, metal prosthesis, etc ...).
* Patient participating or having participated in another clinical study within the last 30 days.
* Patient deprived of liberty following a judicial or administrative decision.
* Patient under guardianship or curatorship.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Negative Biopsy Rate in the treated area | Between 6 to 12 months after treatment

SECONDARY OUTCOMES:
Evaluation of positive biopsy rate in the untreated areas | Between 6 to 12 months after treatment
Rate of side effects | At 12 and 24 months after treatment
Prostate Specific Antigen (PSA) level evolution after treatment | 24 months
Prostate Symptoms | 1 and 2 years(s)
  International Prostate Symptoms Score (IPSS) questionnaire
Continence | 1 and 2 years(s)
  International Continence Society (ICS) questionnaire
Erectile Function | 1 and 2 years(s)
  International Index Erectile Function (IIEF-5) questionnaire
Quality of life | 1 and 2 years(s)
  European Organization for Research and Treatment Quality of Life Questionnaire C30 (EORTC QLQ-C30) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon, France